CLINICAL TRIAL: NCT00311870
Title: Renoprotective Effect of Nisoldipine and Lisinopril in Type 1 Diabetic Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA 92126
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2006-04-06 (Estimated); Status verified 1999-04

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Nisoldipine; Lisinopril

INTERVENTIONS:
Drug: nisoldipine
Drug: lisinopril

SUMMARY:
The aim of the study was to compare the renoprotective effect of a long acting calcium antagonist (nisoldipine) with an angiotensin converting enzyme inhibitor (lisinopril)in type 1 diabetic patients with diabetic kidney disease. In total, 51 patients were randomised to treatment with one of these drugs for 4 years. Changes in kidney function, blood pressure and urinary excretion of albumin were measured every 6 months

ELIGIBILITY:
Inclusion Criteria:

* diabetic nephropathy, type 1 diabetes, hypertension

Exclusion Criteria:

* child bearing potential, non-diabetic kidney disease, malignancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52
Dates: Start 1993-03; Study Completion 1999-04

PRIMARY OUTCOMES:
change in glomerular filtration rate from study start to study end

SECONDARY OUTCOMES:
blood pressure response
change in urinary albumin excretion rate

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, MD, Principal Investigator — Steno Diabetes Center Copenhagen; Hans-Henrik Parving, MD, Study Chair — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Result] Tarnow L, Rossing P, Jensen C, Hansen BV, Parving HH. Long-term renoprotective effect of nisoldipine and lisinopril in type 1 diabetic patients with diabetic nephropathy. Diabetes Care. 2000 Dec;23(12):1725-30. doi: 10.2337/diacare.23.12.1725. PMID 11128341